CLINICAL TRIAL: NCT04305743
Title: Post-procedural Pain Associated With 5 Versus 20 Intravesical Injections of Onabotulinumtoxin A for Treatment of Overactive Bladder: a Multi-center Randomized Controlled Trial
Brief Title: Post-procedural Pain Associated With 5 Versus 20 Intravesical Injections of Onabotulinumtoxin A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Eric Chang, Fellow Physician, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00039851
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Urinary Bladder, Overactive; Incontinence, Urge; Incontinence, Urinary; Urinary Urge Incontinence; Urinary Frequency More Than Once at Night; Nocturia
Keywords: overactive bladder; urgency urinary incontinence; onabotulinumtoxin; bladder; botox
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence; Nocturia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized controlled trial
Who Masked: Participant
Masking Description: Participants are randomized into one of two treatment arms (receiving 5 versus 20 injections per treatment with intradetrusor onabotulinumtoxin A) and are not notified of which arm they are participating in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 Injections (Experimental): Participant's bladder is backfilled with 50 mL of 1% lidocaine for 15 minutes, then drained prior to procedure start. Dose of 100 units onabotulinumtoxin A with dilution to 100 Units/10 mL with preservative-free 0.9% Sodium Chloride Injection is prepared. Cystoscopy is performed. The 23 gauge Laborie InjeTAK needle is inserted 3 mm into the detrusor. 5 injections of 2 mL each (total volume of 10 mL) in a single procedure is performed 1 cm apart in the bladder body. For the final injection, approximately 1 mL of sterile normal saline should be injected such that the remaining onabotulinumtoxin A in the needle is delivered to the bladder.
  Interventions: Drug: OnabotulinumtoxinA 100 UNT
- 20 Injections (Active Comparator): Participant's bladder is backfilled with 50 mL of 1% lidocaine for 15 minutes, then drained prior to procedure start. Dose of 100 units onabotulinumtoxin A with dilution to 100 Units/10 mL with preservative-free 0.9% Sodium Chloride Injection is prepared. Cystoscopy is performed. The 23 gauge Laborie InjeTAK needle is inserted 3 mm into the detrusor. 20 injections of 0.5 mL each (total volume of 10 mL) in a single procedure is performed 1 cm apart in the bladder body. For the final injection, approximately 1 mL of sterile normal saline should be injected such that the remaining onabotulinumtoxin A in the needle is delivered to the bladder.
  Interventions: Drug: OnabotulinumtoxinA 100 UNT

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100 UNT — Intradetrusor onabotulinumtoxin A is administered cystoscopically with 100 unit dose given as either 5 or 20 injections in a single procedure based on the arm the participant is randomized into.
  Other Names: BOTOX

SUMMARY:
Currently, in clinical practice there has been no standardization in the number of injections a single dose of intradetrusor onabotulinumtoxin A is administered in. Given the increasing use of this treatment modality, the aim of this study is to compare outcomes for patients given a 100 unit dose of onabotulinumtoxin A split into 5 as compared to 20 injections for the treatment of overactive bladder or urgency urinary incontinence refractory to medical treatment.

DETAILED DESCRIPTION:
The intradetrusor injection of onabotulinumtoxin A for treatment of idiopathic overactive bladder and urgency urinary incontinence refractory to anticholinergic or β-agonist treatment was approved by the United States Food and Drug Administration (FDA) in 2013. Since then, multiple randomized placebo-controlled trials have demonstrated the effectiveness of the treatment. Currently, Allergan, Inc. and the FDA recommend the intravesical administration of onabotulinumtoxin A with dilution to 100 units/10 mL with preservative-free 0.9% Sodium Chloride Injection, as 20 injections of 0.5 mL each. Currently, in clinical practice there has been no standardization in the number of intravesical injections, with a single dose of onabotulinumtoxin A being administered in as few as 1 injection to as many as 40 injections into the detrusor muscle. Given the increasing use of this treatment modality, the investigators aim to compare patient outcomes for patients given a 100 unit dose of onabotulinumtoxin A split into 5 as compared to the recommended 20 injections for the treatment of idiopathic overactive bladder or urgency urinary incontinence refractory to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women >=18 years of age with diagnosis of urinary urgency, urinary frequency, urgency urinary incontinence, overactive bladder.
* Procedure scheduled in either the outpatient clinic or the operating room to be performed without use of sedation, general, or neuraxial anesthesia.

Exclusion Criteria:

* Male gender.
* Women <18 years of age.
* Non-English speaking.
* Pregnancy (patient will self-report pregnancy).
* Participant has symptoms of overactive bladder due to any known neurological reason (e.g. spinal cord injury, multiple sclerosis, cerebrovascular accident, Alzheimer's disease, Parkinson's disease, etc.)
* Participant uses clean intermittent catheterization or indwelling catheter to manage urinary incontinence.
* Participant has a history or current diagnosis of bladder cancer or other urothelial malignancy.
* Participant has a known allergy or sensitivity to any botulinum toxin preparation.
* Participant has any medical condition that may put her at increased risk with exposure to onabotulinumtoxin A, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis.
* Participant is scheduled for administration of onabotulinumtoxin A with use of sedation, general, or neuraxial anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain from procedure: score | Within 5 minutes of procedure completion
  Pain score as rated on a 10-point visual analog scale within 5 minutes of procedure completion

SECONDARY OUTCOMES:
Duration of procedure | Procedure time
  Total time of procedure defined as time cystoscope is introduced into the bladder to the time the cystoscope is removed from the bladder after completion of all injections
Positive treatment response | 6 weeks post-procedure
  The percentage of patients with a positive treatment response based on answering a Global Response Assessment given 6 weeks after completion of procedure
Urinary tract infections | 12 weeks post-procedure
  Percentage of patients with culture-proven post-procedure urinary tract infections within 12 weeks of procedure
Urinary retention | 12 weeks post-procedure
  Percentage of patients with post-procedure urinary retention requiring clean intermittent catheterization within 12 weeks of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Chang, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of South Florida Health South Tampa Center for Advanced Healthcare, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
All statistical analyses will be performed at the University of South Florida. The investigators performing review of data and statistical analyses will not require the use of, or have access to any personally identifying patient information from either the primary or secondary site of the study.

REFERENCES:
- [Derived] Chang ES, Ringel N, Woodburn KL, Tanner JP, Bassaly R, Greene K, Wyman A, Iglesia C. Postprocedural Pain Associated With 5 Versus 20 Intradetrusor Injections of onabotulinumtoxinA for Treatment of Overactive Bladder: A Multicenter Randomized Clinical Trial. Urogynecology (Phila). 2022 Aug 1;28(8):518-525. doi: 10.1097/SPV.0000000000001199. Epub 2022 May 12. PMID 35543540